CLINICAL TRIAL: NCT04061889
Title: Clinical Epidemiology Cohort Study for Patient Living With HIV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Hung Chin Tsai, Visiting Physician, Kaohsiung Veterans General Hospital.
Other Study IDs: VGHKS19-CT4-02
Record Dates: First submitted 2019-08-15; First posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: intervention name is not applicable — Another intervention is not applicable either, due to the observational study design

SUMMARY:
This is a retrospective observational cohort study for the patient living with HIV aiming to understand more in disease progress, resistant mutation, comorbidity, and common coinfection.

ELIGIBILITY:
Inclusion Criteria:

* Patient living with HIV receiving follow-up in Kaohsiung VGH

Exclusion Criteria:

* not applicable

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1 infected adult
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Hazard ratio of cohort epidemiology characteristics in treatment failure, renal failure and hepatitis D coinfection | on average of 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Hung Chin Tsai, MD,PhD, Study Chair — Kaohsiung Veteran General Hospital
Locations (1):
- Kaohsiung Veteran General Hospital, Kaohsiung City, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided